CLINICAL TRIAL: NCT00346879
Title: Thromboprophylaxis in the Morbidly Obese With Weight Based Dosing of Fondaparinux: A Pharmacodynamic Study
Brief Title: Study to Determine Effective Dosing of Fondaparinux in Obese Persons
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn; study closed due to lack of accrual.
Sponsor: Indiana University School of Medicine (Other)
Collaborators: American Society for Bariatric Surgery (Other)
Responsible Party: Samer Mattar, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0602-26
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity
Keywords: fondaparinux for prevention of blood clots
MeSH Terms: conditions — Obesity, Morbid | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fondaparinux — Single 2.5 mg dose of fondaparinux or weight-based 0.03 mg/Kg dose of fondaparinux

SUMMARY:
This is a prospective open-label study comparing two dosing regimens of fondaparinux, which is used to prevent deep vein thrombosis, in morbidly obese volunteers.

DETAILED DESCRIPTION:
The incidence of obesity is growing at an alarming pace and has reached epidemic proportions. Subjects who are more than 100 pounds over their ideal body weight are classified as being morbidly obese and are considered to carry a high risk for multiple chronic medical conditions that impact quality of life and shorten life span. As a result of obesity, these individuals are also at a higher risk for developing life-threatening blood clots. Such risk is further elevated with exposure of obese subjects to the stress of surgery. In fact, the most common cause of death after major surgery in morbidly obese subjects is the migration of blood clots to the lung and heart. With the current rise in popularity of weight loss surgery, it has become imperative that we identify a medication that is safe and effective in preventing the formation of blood clots. Fondaparinux has the potential for being an effective anti-clotting drug. It is superior to other similar drugs because it is completely utilized by the body, and has a more predictable action. The problem, however, is that the recommended doses for fondaparinux were obtained after studies on lean individuals. This is a fixed dose that is administered universally, regardless of the size of the subject. Presently, we have no information on what the recommended doses should be for morbidly obese subjects, who are in the most need for effective anti-clotting medication. This study will attempt to determine whether a fixed dose or a weight-related dose is appropriate for morbidly obese subjects, and also investigate the safety of administering weight-based dosing to these individuals.

ELIGIBILITY:
Inclusion Criteria:

- Age 19-65 BMI: 35-65 Negative pregnancy test on day of study

Exclusion Criteria:

- Blood Pressure < or = to 160/90 Temperature > 37.5 C (99.5 F) Nursing a baby Positive pregnancy test on day of study. Medications: History of regular treatment with anticoagulants or any anti-platelet agents including aspirin and other NSAIDS; use of aspirin or other NSAIDS within 1 month of study.

Past Medical History:

Cerebrovascular accident (including transient ischemic attacks) within 6 months of study.

Diabetic retinopathy as documented by positive fundoscopy in previous 3 months. Active peptic ulcer disease, by EGD or Ba meal, within 3 months of study. Known bleeding disorder. Known thrombophilia History of heparin induced thrombocytopenia. History of bacterial endocarditis. Known hypersensitivity to fondaparinux. Ulcerative colitis. History of GI bleeding History of hematuria Recent surgery (in previous 3 months). Recent trauma - road traffic accident (previous 3 months).

Laboratory Values:

Platelet count < or = to 100,000. Hemoglobin <12g/dl - women or <14g/dl - men. Prothrombin time > 13s Activated partial thromboplastin time (APTT) > 35s Liver function test parameters: ALT > 60u/L, AST > 40u/L, γ-GT >85u/L, Alkaline phosphatase >251 u/L or total bilirubin > 1.3 mg/dl.

Estimated urinary creatinine clearance < 50 mls/min. Hematuria on urine dipstick.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Compare peak anti-Xa activity between fixed dose and weight-based dose of fondaparinux | 5 days

SECONDARY OUTCOMES:
Determine safety of fondaparinux in the two treatment groups | 5 days
Determine if anti-Xa activity accumulates | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Samer Mattar, MD, Principal Investigator — Indiana University
Locations (1):
- Clarian Bariatric Center, Indianapolis, Indiana, United States